CLINICAL TRIAL: NCT07378111
Title: Acceptability (Including Gastrointestinal Tolerance, Compliance) of a Vegetarian Paediatric Enteral Tube Feed With Food Derived Ingredients.
Brief Title: Vegetarian Tube Feed Study
Acronym: Tube feed
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPV tube feed PB002; IRAS ID 341165 (Other: Yorkshire & The Humber - South Yorkshire Research Ethics Committee)
Record Dates: First submitted 2026-01-08; First posted 2026-01-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Paediatric

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children will act as their own control for the nutritional product (Experimental): Gastrointestinal tolerance and daily formula intake over 28 days.
  Interventions: Dietary Supplement: paediatric tube feed

INTERVENTIONS:
Dietary Supplement: paediatric tube feed — 500ml tube feed to be provided daily over 28 days.

SUMMARY:
This is a single arm, prospective, single-centre study to evaluate the gastrointestinal tolerance and compliance over a 28-day period using a tube feed with food derived ingredients.

DETAILED DESCRIPTION:
Acceptability (including gastrointestinal tolerance, compliance of a paediatric vegetarian tube feed with food derived ingredients. Gastrointestinal tolerance will data will be collected using a 4point Likert scale, daily record of tube feed volume intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 1 -15 years requiring more than 50% of energy from tube feeding or to take alongside home-made blended diet as part of their dietary management for disease related malnutrition.
* Patients well-established and stable on current nutritional support regimen. Willingly given, written, informed consent from patient/caregiver

Exclusion Criteria:

* No established tube feed.
* Inability to comply with the study protocol, in the opinion of the investigator.
* Under 1 years of age
* Patients on parenteral nutrition
* Known food allergies, including to any ingredients listed in appendix 1.
* Participation in another interventional study within 2 weeks of this study.
* Patients with known or suspected ileus or mechanical bowel obstruction

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal tolerance and formula intake | From enrolment to end of study over 28 days
  Daily gastrointestinal tolerance measured using a 4 point Likert scale of none, mild, moderate, severe symptoms over days.
Formula volume intake in mL | From enrolment to end of study over 28 days
  Formula intake measured daily in mLs over 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Graeme O'Connor, PHD, Principal Investigator — Great Ormond Street Hospital Nutrition and Dietetics Department

IPD SHARING:
Plan to Share IPD: No